CLINICAL TRIAL: NCT03293602
Title: MISOBOLD - Prostate Cancer Hypoxia Using BOLD MRI and 18F-MISO PET Imagin
Brief Title: MISOBOLD - Prostate Cancer Hypoxia Using BOLD MRI and 18F-MISO PET Imaging
Acronym: MISOBOLD
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: the team has changed. the new team did not have the perosnnel to set up the study
Sponsor: University Hospital, Bordeaux (Other)
Collaborators: Cancéropôle GSO and GIRCI SOOM (API-K) (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CHUBX 2014/26
Record Dates: First submitted 2017-09-20; First posted 2017-09-26 (Actual); Last update posted 2019-11-27 (Actual); Status verified 2019-11

CONDITIONS: Prostate Cancer
Keywords: prostate cancer; MRI; BOLD; 18F-MISO; PET
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- F-MISO PET imaging (Experimental): F-MISO PET imaging will be added to the preoperative staging explorations of a patient with high risk prostate cancer candidate to radical prostatectomy. Patient will be selected during multidisciplinary meeting and urology consultation of Bordeaux and Toulouse university hospitals. Functional MRI imaging should be available before surgery. If patient consent to participate in the study, F-MISO PET imaging will be planed before prostatectomy. Results of this exam will not be considered for patient therapeutic management.
  Interventions: Device: F-MISO PET imaging

INTERVENTIONS:
Device: F-MISO PET imaging — F-MISO PET imaging will be added to the preoperative staging explorations of a patient with high risk prostate cancer candidate to radical prostatectomy. Patient will be selected during multidisciplinary meeting and urology consultation of Bordeaux and Toulouse university hospitals. Functional MRI imaging should be available before surgery. If patient consent to participate in the study, F-MISO PET imaging will be planed before prostatectomy. Results of this exam will not be considered for patient therapeutic management.

SUMMARY:
This feasibility exploratory study objective is to assess the ability of combined MRI BOLD and 18F-MISO PET imaging to visualize tumor hypoxia compare to histological results obtained after radical prostatectomy in order to, in time, be able to identify patient with bad prognostic and to offer them the best therapeutic strategy.

DETAILED DESCRIPTION:
Prostate cancer is the fisrt one in male with 80.000 new cases each year in France. Forty thousand curative treatments are performed each year, but 25 to 30% of these patients will present a cancer reccurence after radical surgery or conformationnal radiotherapy, Tissu hypoxia seems to be mainly responsible of the local reccurence and conduct to molecular damages that creates carcinogenesis and tumor agressitivity. This hypoxia inhibits the DNA healing and the apoptosis but increases the angiogenesis, that leads to treatment resistance. L. Marignol &al clearly showed that hypoxia may have a main role in hormonal resistance. Furthermore, M. Milosevic & al showed that hypoxia is an independent factor of local reccurence after radiotherapy. Nowadays, new technics of IMRT in radiotherapy planning could be able to target an hypoxic prostate region to prevent reccurence. Patients who are eligible to radical prostatectomy will benefit of a prostate MRI with BOLD sequences and a 18F-misonidazole PET before surgery. The results of these two technics will be compared to the histological results using CAIX and HIF immunohistochemistery markers

ELIGIBILITY:
Inclusion Criteria:

* Patient above 18.
* Prostate tumor with histological confirmed diagnosis and highly radiological suspected target on MRI
* High risk patient : >T2c grade, Glasgow score > 7 and PSA > 20ng/ml
* Surgical treatment chosen during multidisciplinary meeting
* ECOG ≤2
* Patient must have undergone MRI with BOLD sequence less than 6 month prior surgery
* Member or beneficiary of a social security system.
* Signed informed consent.

Exclusion Criteria:

* Patient included in another clinical study
* Geographical, social or psychological reasons preventing patient from submitting to the study's medical monitoring
* Patient deprive of liberty, adult subjects to legal protection or unable to give consent
* Contraindications to MRI
* Contraindication to gadolinium injection

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-09-01 (Estimated); Primary Completion 2020-01-01 (Estimated); Study Completion 2020-01-01 (Estimated)

PRIMARY OUTCOMES:
comparison between histological results and oxygenation quantitative values from MRI and PET exams | Inclusion, 1 month
  Correlation study between anatomopatology data, product by prostatectomy anatomic piece, using HIF1-CAIX histological markers and:
  * on one hand PET FMISO uptake
  * on the other hand, MRI BOLD signal

SECONDARY OUTCOMES:
quantitative analysis | Inclusion, 1 month
  a quantitative analysis of inter-individual variability will be done in order o compare inter-individual variability of hypoxia measures between the two imaging modalities

CONTACTS AND LOCATIONS:
Locations (1):
- Centre de Lutte Contre le Cancer, Toulouse, France

IPD SHARING:
Plan to Share IPD: No